## A Novel Neuromonitoring Guided Cognitive Intervention for Targeted Enhancement of Working Memory

Statistical Analysis Plan

NCT04002167

August 25, 2023

The statistical analysis was computed in RStudio (R version 4.3.0) and the linear mixed-effect models for each behavioral dataset were constructed in Imer package to handle the missing date points. The analysis incorporated the interaction between group and session as a fixed effect, accounting for age, sex, and medication effects, while subject IDs were treated as a random effect in the model.